CLINICAL TRIAL: NCT06221072
Title: A Phase III, Multicenter, Randomized, Double-blind Clinical Trail to Assess JMT103 Compared to Azoledronic Acid for the Prevention of Bone-related Events in Patients With Bone Metastases From Malignant Solid Tumors
Brief Title: A Study to Assess the Prevention of Bone-related Events in Patients With Bone Metastases From Malignant Solid Tumors Treated With JMT103 Compared to Zoledronic Acid
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JMT103-012
Record Dates: First submitted 2024-01-14; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Imaging Examination Shows at Least One Site With Bone Metastases From Soild Tumors
MeSH Terms: interventions — Zoledronic Acid

STUDY DESIGN:
Intervention Model Description: multicenter, randomized, double-blind clinical Trail
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1-JMT103 (Experimental): Participants will receive JMT103 and zoledronic acid placebo.
  Interventions: Drug: JMT103
- Group 2-zoledronic acid (Experimental): Participants will receive zoledronic acid and JMT103 placebo.
  Interventions: Drug: zoledronic acid

INTERVENTIONS:
Drug: JMT103 — 120 mg by subcutaneous injection every 4 weeks
  Arms: Group 1-JMT103
Drug: zoledronic acid — 4 mg by intravenous drip (100mL:4mg) every 4 weeks
  Arms: Group 2-zoledronic acid

SUMMARY:
This is a phase Ⅲ, multicenter, randomized, double-blind, study to evaluate the efficacy and safety of JMT103 in patients with bone metastases from malignant solid tumors. The purpose of this study is to determine if JMT103 is non-inferior to zoledronic acid.

ELIGIBILITY:
Inclusion Criteria:

1. Age: older than 18 years;
2. Breast cancer, prostate cancer, lung cancer and other solid tumors diagnosed by histological or cytological examination (prostate patients should also meet: castration-resistant prostate cancer with serum testosterone <50 ng/dL or 1.7 nmol/L and serum PSA progression after surgery or drug castration treatment);
3. Patients with imaging studies showing at least one tumor bone metastasis;
4. With a good organ function;
5. Expected survival of at least 6 months.

Exclusion Criteria:

1. Previous or ongoing osteomyelitis or osteonecrosis of the jaw; dental or oral surgery; acute dental or jaw disease requiring oral surgery; invasive dental procedures planned during the study; patients with pulpitis during the screening period;
2. Radiotherapy or surgery for the bone metastases is planned during the study;
3. Patients with brain metastasis or meningeal metastasis (patients with neurological symptoms should undergo MRI/CT examination to exclude patients with brain metastasis);
4. Patients with bone metabolic diseases [e.g., Paget's disease, Cushing's syndrome, hyperprolactinemia, hyperthyroidism/hypothyroid (except for hypothyroidism with normal TSH, FT3, and FT4 after stable thyroid hormone replacement therapy, and subclinical hypothyroidism that does not need to be treated), hyper/hypoparathyroidism, etc.];
5. Uncontrolled concurrent diseases, including but not limited to: uncontrolled diabetes mellitus (≥grade 3, NCI-CTCAE 5.0), symptomatic congestive heart failure, hypertension (BP> 150/90 mmHg after standard therapy), unstable angina, arrhythmia requiring medical or instrumental treatment, history of myocardial infarction within 6 months, echocardiography with left ventricular ejection fraction <50%;
6. Treatment with anti-RANKL antibody, bisphosphonates (except for bone scan purposes) within 6 months prior to the first dose;
7. Patients considered by the investigator as unsuitable for this study (such as poor compliance, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1360 (Estimated)
Dates: Start 2024-04-05 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Time to the First on-study Skeletal-Related Event (SRE) | Up to approximately 48 months

SECONDARY OUTCOMES:
Time to First and Subsequent SRE (21 days from the last SRE is subsequent SRE) | Up to approximately 48 months
Percent change from baseline in Urinary N-Telopeptide Corrected for Urine Creatinine (NTx/Cr) | Up to approximately 28 months
Quality of life score (concise pain assessment Scale and EQ-5D-5L scale); | Up to approximately 48 months
Incidence and severity of adverse events (AEs) | Up to approximately 48 months
JMT103 The incidence of injection anti-drug antibodies (ADA) and neutralizing antibodies (Nab) | Up to approximately 48 months
Serum concentration of JMT103 | Up to approximately 48 months
Overall survival (OS) | Up to approximately 6 years

IPD SHARING:
Plan to Share IPD: No